CLINICAL TRIAL: NCT02342197
Title: Comparative Study Between Minidose Long Protocol and Microdose Flare Protocol in Controlled Ovarian Hyperstimulation for Poor Responders in ICSI Cycles
Brief Title: Comparative Study Between Minidose Long Protocol and Microdose Flare Protocol in Controlled Ovarian Hyperstimulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Nawara Mohamed Hashish, Nawara Hashish, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 610012011
Record Dates: First submitted 2014-12-28; First posted 2015-01-19 (Estimated); Results first posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
Keywords: Low responders; Minidose long protocol; Microdose flare protocol; Oocyte yield
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minidose long protocol (Active Comparator): Half dose of GnRH agonist (Decapeptyl 0.05) was started in the midluteal phase and Gn's was started from the second day of the cycle.
  Interventions: Drug: Decapeptyl
- Microdose flare protocol (Active Comparator): Half the dose of GnRH agonist (Decapeptyl 0.05) was started on the second day of the cycle together with Gn's
  Interventions: Drug: Decapeptyl

INTERVENTIONS:
Drug: Decapeptyl — half the dose of Gn agonist
  Other Names: GnRH agonist

SUMMARY:
Objective: To compare two stimulation protocols, the minidose long protocol and the microdose flare protocol designed for low responders undergoing ICSI.

Design: Randomized prospective study. Setting: University hospital IVF unit. Patients: 60 poor responder patients coming for IVF center for ICSI. Interventions: Minidose long protocol in which half the dose of agonist was administered from the mid luteal phase until the day of HCG administration was compared with microdose flare protocol in which half the dose of GnRH was administered from the second day of the cycle until the day of HCG administration. Both groups received Gn stimulation from the second day of the cycle (300-450 IU).

Main outcome measures: Number of oocytes retrieved.

DETAILED DESCRIPTION:
Patients and methods:

60 patients expected to have poor response for ovarian stimulation attending kasr EL-Aini hospital IVF center planning for ICSI during the year 2011 were randomized to receive ovulation induction for controlled ovarian hyperstimulation by either one of two protocols: Minidose long protocol and microdose flare protocol.

Inclusion criteria:

All patients included were classified as poor responders when one of the following criteria was present:

* Age > 35 years.
* Day 3 serum FSH level > 10m IU/ml.
* Number of antral follicles measuring 4-8mm during the early phase < 6.
* Small ovarian volume.
* AMH < 1.
* Prior poor ovarian response to COH (oocytes < 5).

Exclusion criteria:

* Polycystic ovarian syndrome patients.
* Patients with Endometriosis.
* Normal responders to ovulation induction.
* Patients having ovarian cyst.
* Patients receiving ovulation induction in the preceding cycle. The study was approved by Kasr El-Aini IVF center research committee. Each patient had given informed consent after full explanation of the procedure. Randomization was performed according to a computer generated list. The patients were randomized to two groups.

The Minidose long protocol:

Decapeptyl 50µg/ day was administered SC from cycle day 21 until menstruation. On the second day of the cycle, patients were assessed for downregulation; E2 level < 50 pg/ml, endometrial thickness less than 5 mm, no follicles > 15mm. Once patient downregulation was confirmed, Gn dose was commenced at an initial dose of 300-450 IU/day for the first 5 days followed by individual adjustment in Gn dose according to ovarian response and the dose of Decapeptyl 50µg/day was continued until day of HCG administration.

The microdose flare protocol:

Administration of OCP's at the prior menses followed by Decapeptyl 50µg/day SC started on the second day of the cycle and continued until the day of HCG administration. Gn was started concomitantly on the second day of the cycle as described above.

Cycle monitoring:

Monitoring consisted of several ultrasound examination and serum E2 level in both protocols. The starting Gn dosage was determined by a combination of factors including patient age, ovarian reserve testing, prior stimulation response and was adjusted according to individual response. Serum LH levels were measured from day 6 of stimulation to exclude premature luteinization (LH > 15 IU/L).

10,000 IU HCG was administered intramuscular when at least two leading follicles were 18mm in diameter. Oocyte retrieval was performed 35 hours after HCG administration by ultrasound guided transvaginal aspiration.

Laboratory procedures:

The ICSI procedure was performed 4 hours after oocyte aspiration for all the mature oocytes. Fertilization was assessed 16-18 hours after ICSI and was considered normal only when two distinct pronuclei were present. The embryos obtained were categorized on day 2-3 into 3 grades depending on their morphological appearance, zonal thickness, cytoplasmic fragmentation and blastomere size.

Transfer procedure and luteal support:

Depending on patient age, embryo quality and the number of embryos available, 1-4 embryos were transferred 2-3 days after oocyte collection under transabdominal ultrasound guidance using a cook catheter.

The luteal phase was supported with micronized progesterone 400 mg twice daily administered vaginally until a pregnancy test was performed.

Outcome measures:

To assess a difference in pregnancy rates between the two protocols, a sample size of 100's of patients should be considered but considering the size of our work, it would be many years before such large samples could be recruited. We therefore chose to focus on oocyte number as a main outcome measure.

The data recorded for analysis included: age, infertility history and etiology, day 3 FSH, duration of stimulation, number of gonadotrophin ampoules required, E2 level on the day of HCG administration, number of oocytes retrieved and fertilized and number of embryos transferred.

The primary outcome measure was the number of oocytes retrieved. The secondary outcome measures were implantation and clinical pregnancy rates. A clinical pregnancy was defined as a normal gestational sac measured with transvaginal ultrasound after 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 35 years
* Day 3 serum FSH level > 10m IU/ml
* Number of antral follicles measuring 4-8mm during the early phase < 6
* Small ovarian volume
* AMH < 1
* Prior poor ovarian response to COH (oocytes < 5)

Exclusion Criteria:

* Polycystic ovarian syndrome patients
* Patients with Endometriosis
* Normal responders to ovulation induction
* Patients having ovarian cyst
* Patients receiving ovulation induction in the preceding cycle

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minidose Long Protocol | Microdose Flare Protocol
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minidose Long Protocol | Microdose Flare Protocol | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (1.5) | 37.1 (1.5) | 37.2 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
BMI (kg/m2) [Mean (Standard Deviation); unit: kg / m2] | 30 (2.5) | 31 (1.8) | 30.5 (0.2)
Day 3 FSH (IU/L) [Mean (Standard Deviation); unit: IU/L] | 8 (1.1) | 7.6 (1.1) | 7.8 (0.1)
Duration of infertility [Mean (Standard Deviation); unit: years] | 5.1 (1.5) | 5.7 (1.5) | 5.4 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Minidose Long Protocol | Microdose Flare Protocol
Number analyzed (Participants) | 27 | 28
oocytes | 4 (1) | 3.4 (0.7)

ADVERSE EVENTS:
Arm/Group | Minidose Long Protocol | Microdose Flare Protocol
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minidose Long Protocol (N=0) | Microdose Flare Protocol (N=0)
ovarian hyperstimulation (Endocrine disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes